CLINICAL TRIAL: NCT04267159
Title: Acute Atrial Fibrillation and Flutter Treated Electively - a Randomized Controlled Clinical Trial on the Safety of Elective Management of Acute Atrial Fibrillation and Flutter
Brief Title: Acute Atrial Fibrillation and Flutter Treated Electively
Acronym: AFFELECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Responsible Party: Principal Investigator, Jussi Hernesniemi, Professor, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETL R19133
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Intervention Model Description: The AFFECT trial is a randomized clinical trial with a non-inferioirity setting studying the applicability of delayed rhythm control in the management of acute paroxysmal or persistent atrial fibrillation or flutter.
  Patients are randomized to two treatment protocols in 2:3 ratio. For every two patients randomized to conventional treatment, three patients are randomized to experimental treatment. The randomization ratio is designed to allow for maximally one third of the patients in the experimental treatment group to drop-out without compromising the power of the study.
  Overall five hundred patients are required to show non-inferiority with a one-sided alpha value 0.025 and 90% power expecting a maximal drop out rate of 33% (n=100) from the experimental treatment arm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional treatment by acute cardioversion (Active Comparator): Participants in the conventional treatment arm will be returned to sinus rhythm in the emergency department within 48 hours of symptom onset unless they convert to sinus rhythm spontaneously.
  Interventions: Other: Acute cardioversion
- Elective treatment by delayed cardioversion (Experimental): Participants in the elective treatment arm will be returned to sinus rhythm in an out-patient clinic approximately one week after randomizatio unless they convert to sinus rhythm spontaneously.
  Interventions: Other: Delayed cardioversion

INTERVENTIONS:
Other: Acute cardioversion — Acute restoration of sinus rhythm by medical or electrical cardioversion in the emergency department
  Arms: Conventional treatment by acute cardioversion
Other: Delayed cardioversion — Delayed restoration of sinus rhythm by medical or electrical cardioversion in the out-patient clinic
  Arms: Elective treatment by delayed cardioversion

SUMMARY:
The AFFELECT -study compares two types of treatment modalities for acute atrial fibrillation or flutter for patients in whom rhythm control is desirable. The main purpose is to observe if these arrhythmias can be safely treated electively (within 5-9 days).

All patients are recruited in the emergency department. Patients must be in good clinical condition so that they can be discharged regardless to which treatment modality is randomly selected to them. Patients randomized to conventional care are treated conventionally which means acute rhythm control is applied by electrical or medical cardioversion in the emergency department (within 48 hours of onset of the arrhythmia). Patients randomized to elective care are discharged immediately after adequate temporary rhythm control is assured.

All patients will visit a cardiologist out-patient clinic at approximately one week after the emergency room visit. Patients randomized to elective treatment and still in atrial fibrillation or in atrial flutter will be restored to sinus rhythm by electrical or medical cardioversion at the out-patient clinic. Cardiovascular status and treatment options are evaluated for all patients.

Anticoagulation is managed according existing guidelines for all patients. Due to possibility of delayed cardioversion in the interventional group (elective care group), all patients receive anticoagulation before the out-patient clinic despite their thromboembolic risk. All patients who have not received adequate anticoagulation for three weeks prior to the delayed cardioversion will undergo a transesophageal cardiac ultrasound to ensure they are not in excess risk for thromboembolic events. Patients randomized to elective treatment have the possibility to opt-out and undergo acute cardioversion if their symptoms are unmanageable during the first week before the out-patient clinical.

All patients are monitored for their symptoms by a standardized quality-of-life questionnaire and for possibly required acute medical interventions during the first week and one month after the out-patient clinic. After one month, all patients undergo an electrocardiography (ECG) to ensure the maintenance of normal rhythm in both treatment groups. After the months follow-up all patients are subsequently monitored for a maximum of five years for need of medical interventions due to atrial fibrillation of atrial flutter. New antiarrhythmics such as flecainide are not prescribed during the first month.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with acute (<48hours) atrial fibrillation or atrial flutter to ER
* Planned acute rhythm control for the arrhythmia by the attending physician in ER
* Good perceived health as assessed by attending physician in ER
* Resting heart rate 110bpm or lower before or after adequate rate control therapy

Exclusion Criteria:

* Haemodynamically stable (mean arterial pressure above 60mmHg)
* Need for acute restoration of sinus rhythm due to some other somatic cause
* No other major complicating acute illness (e.g. decompensated HF or acute MI)
* Anticoagulation not safe
* Mechanical heart valve or mitral stenosis
* The need for prolonged (>24h) hospitalization due to any cause
* Exceptionally high risk for thromboembolic events (e.g. history of thromboembolic stroke regardless of adequate anticoagulation)
* Transesophageal echocardiography contraindicated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Sinus Rhythm | One month after preplanned out-patient clinic visit
  Prevalence of sinus rhythm in the treatment arms measured by electrocardiography

SECONDARY OUTCOMES:
Number of cardioversions after emergency department | First week after randomization and before the preplanned out-patient clinic
  The number of performed cardioversions (electrical or medical)
Number of cardioversions after out-patient clinic | One month after out-patient clinic
  The number of performed cardioversions (electrical or medical)
Overall number of cardioversions | From randomization to the end of first month follow-up after out-patient clinic visit
  The number of performed cardioversions (electrical or medical)
Drop-out from delayed cardioversion group | Four days or earlier after randomization to elective (delayed) treatment group
  The number of subjects needing unplanned cardioversion before preplanned out-patient clinic visit (four days or earlier after randomization) due to medical reasons or due to subjectively perceived unbearable symptoms (EHRA III or IV).
Rehospitalization due to cardiovascular causes | One week before and one month after out-patient clinic visit
  Rehospitalization due to any cardiovascular cause
Immediate quality of life | First week after randomization and before the preplanned out-patient clinic
  Quality of life as assessed by questionnaires depicting quality of life (AFEQT)
Quality of life after out-patient clinic | One month after out-patient clinic
  Quality of life as assessed by questionnaires depicting quality of life (AFEQT)

CONTACTS AND LOCATIONS:
Overall Officials: Jussi A Hernesniemi, MD, PhD, Principal Investigator — TAYS Heart Hospital and Tampere University
Locations (4):
- Finland (4):
  - Central Finland Central Hospital, Jyväskylä, Central Finland
  - Kanta-Häme Central Hospital, Hämeenlinna, Kanta-Häme
  - Päijät-Häme Central Hospital, Lahti, Paijat-Hame Region
  - Tampere University Hospital, Tampere, Pirkanmaa

IPD SHARING:
Plan to Share IPD: No
IPD can be shared only upon reasonable request after full anonymization by the discretion of the study review board.